CLINICAL TRIAL: NCT02879006
Title: Double-Blind, Placebo-Controlled Phase 2 Study to Assess Safety and Efficacy of Chinese Herbal Therapy and Multiple Food Allergen Oral Immunotherapy
Brief Title: E-B-FAHF-2, Multi OIT and Xolair (Omalizumab) for Food Allergy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiu-Min Li (Other)
Responsible Party: Sponsor-Investigator, Xiu-Min Li, Professorial Lecturer, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 16-1384
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Food Allergy
Keywords: Chinese herbal therapy; Oral immunotherapy; Food allergy; Omalizumab
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese Herbal Medication (Active Comparator)
  Interventions: Drug: Chinese Herbal Medication; Drug: Omalizumab; Drug: Multi OIT
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Omalizumab; Drug: Multi OIT

INTERVENTIONS:
Drug: Chinese Herbal Medication — Capsules, 26 month course, starting 2 months pre-OIT
  Other Names: E-B-FAHF-2
  Arms: Chinese Herbal Medication
Drug: Placebo — Placebo capsules that look identical to E-B-FAHF-2, 26 month course, starting 2 months pre-OIT
  Other Names: Placebo Chinese Herb
  Arms: Placebo
Drug: Omalizumab — 4 months course, starting 2 months pre-OIT through the 2 month build-up phase
  Other Names: Xolair®
Drug: Multi OIT — 24 months of multi OIT (maintenance dose of 1gm each food allergen)

SUMMARY:
The purpose of this study is testing the use E-B-FAHF-2 Chinese herbal therapy in combination with multi-food oral immunotherapy (OIT) and Xolair® (Omalizumab) to help children and adults who are allergic to foods be able to safely tolerate food allergens. Specifically in this protocol, the food allergens are milk, egg, peanut, almond, cashew, hazelnut, walnut, sesame, and/or wheat. Omalizumab is considered an investigational drug for the treatment of food allergies in children and adults. Investigational means it has not been approved by the Food and Drug Administration (FDA) for use in the U.S. The researchers hope to learn whether the addition of Chinese herbal therapy (E-B-FAHF-2) can improve the outcome of sustained unresponsiveness (which is the ability to consume a food allergen and pass an oral food challenge after being off treatment for 3 months) as compared to placebo (i.e. subjects with OIT/Omalizumab + herbal vs. OIT/Omalizumab + placebo), and will help adults and children be able to safely ingest the foods they are allergic to.

DETAILED DESCRIPTION:
Prior studies have shown that this Chinese herbal formulation is safe and well-tolerated in food allergic individuals. While oral immunotherapy (OIT) can lead to desensitization, it remains uncertain whether this treatment can lead to lasting protection. Therefore, this study aims to use the Chinese herbal formula in combination with OIT to determine whether sustained protection can be achieved. All subjects will receive multi-allergen OIT, along with a 4 month course of omalizumab to provide added safety for the initial dose escalation and build up phases. Subjects will be randomized to receive active Chinese herbal formula or placebo. Subjects will be treated with OIT for 2 years and then food challenges will be performed to assess for desensitization. For those who achieve desensitization, all treatments will be discontinued and food challenges will be performed 3 months later to assess for sustained unresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* 6 through 40 years
* At least one of the following for each of the 3 study allergens: serum IgE >4 kU/L or skin prick test >6mm
* dose limiting symptoms at a cumulative dose of <=444 mg protein for 3 allergens as screening double-blind, placebo-controlled food challenge
* use of an effective method of contraception by females of child-bearing potential
* ability to ingest oat or corn with no allergic reaction

Exclusion Criteria:

* If baked milk or egg are tolerated (assessed by clinical report), then milk or egg may not be included as a study allergen
* Any disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, and serious ventricular arrhythmias
* History of other chronic disease requiring therapy (other than asthma, atopic dermatitis, or rhinitis)
* History of eosinophilic gastrointestinal disease
* Current participation in any other interventional study
* Investigational drug use within 90 days
* Subject is on build-up phase of any allergen immunotherapy (prior to maintenance dosing)
* Current uncontrolled moderate to severe asthma as defined by:

  * FEV1 value <80% predicted (or PFR if unable to perform spirometry) or any clinical features of moderate or severe persistent asthma baseline severity (as defined by the 2007 NHLBI Guidelines) and greater than high daily doses of inhaled corticosteroids (as defined for children and adults using dosing tables from the 2007 NHLBI Guidelines).
  * Use of steroid medications in the following manners: history of daily oral steroid dosing for >1 month during the past year, having 1 burst or steroid course within the past 6 months, or having >1 burst oral steroid course within the past 12 months.
  * Asthma requiring >1 hospitalization in the past year for asthma or >1 ED visit in the past 6 months for asthma.
* Use of systemic steroid medications (IV, IM or oral) for indications other than asthma for > 3 weeks within the past 6 months
* Inability to discontinue antihistamines for the initial day of escalation, skin testing or DBPCFC
* Use of Xolair® (omalizumab) within the past 6 months
* Known sensitivity to Xolair® (omalizumab) or to the class of study drugs
* Body weight more than 90 kg, or subjects with weight-IgE combination that yields a dose requirement greater than 600 mg dosing
* Use of beta-blockers (oral), (ACE) inhibitors, angiotensin-receptor blockers or calcium channel blockers
* Pregnancy or lactation
* Inability to swallow placebo capsules
* Mental illness or history of drug or alcohol abuse that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements

Ages: 6 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2016-08; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Sustained unresponsiveness | month 29
  Sustained unresponsiveness evaluated by the absence of dose-limiting symptoms to a cumulative dose of 4,444 protein.

SECONDARY OUTCOMES:
Desensitizing to 4444mg | month 26
  Number of participants tolerating a cumulative dose of 4,444mg of food allergen protein.
High level of desensitization to 7444mg or higher | month 26
  Number of participants tolerating a cumulative dose of 7,444mg or higher (max of 10,444mg) of food allergen protein

CONTACTS AND LOCATIONS:
Overall Officials: Julie Wang, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Wang ZZ, Geliebter J, Tiwari R, Li XM. Traditional Chinese medicine for food allergy and eczema. Ann Allergy Asthma Immunol. 2021 Jun;126(6):639-654. doi: 10.1016/j.anai.2020.12.002. Epub 2020 Dec 10. PMID 33310179